CLINICAL TRIAL: NCT06925698
Title: Immunosuppressive Therapy Alone Versus Immunosuppressive Therapy Plus Oral Anticoagulation in the Treatment of Lower Extremity Venous Thrombosis Associated With Behcet's Disease
Brief Title: Immunosuppressive Therapy Alone Versus Plus Oral Anticoagulation in the Treatment of VT Associated With Behcet's Disease
Acronym: BETTER
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Marmara University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09.2023.1733
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Behcet Disease; Behcet Disease and Vascular Involvement; Deep Venous Thromboses; Post Thrombotic Syndrome
Keywords: Behcet's disease; Deep venous thrombosis; Anticoagulant therapy; Rivaroxaban
MeSH Terms: conditions — Behcet Syndrome; Venous Thrombosis; Postthrombotic Syndrome | interventions — Immunosuppression Therapy; Rivaroxaban; Immune Tolerance

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective, randomized, double-blind, placebo-controlled, Phase III clinical trial designed to evaluate the efficacy and safety of immunosuppressive therapy alone versus immunosuppressive therapy plus oral anticoagulation (Rivaroxaban) in the treatment of venous thrombosis associated with Behçet's Disease.
  Participants will be randomized (1:1) into two groups:
  Immunosuppressive therapy alone Immunosuppressive therapy plus Rivaroxaban (20 mg/day, oral) The treatment duration is 12 months, with follow-up visits at weeks 2, 4, months 2, 3, 6, 9, and 12.
  The study employs a double-blind design, meaning that both participants and investigators are blinded to treatment allocation. Randomization is stratified by gender to ensure balanced distribution.
  The primary endpoint is the rate of thrombotic relapse within 52 weeks, assessed via venous Doppler ultrasound. Secondary outcomes include post-thrombotic syndrome development, quality of life measures, and safety ass
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study follows a double-blind design, ensuring that participants, care providers, investigators, and outcomes assessors are all blinded to the treatment allocation. Randomization and treatment assignment are managed by an independent data monitoring team, which is also responsible for ensuring the integrity of the blinding process.
  The placebo and active treatment (Rivaroxaban) are identical in appearance, dosage, and administration, minimizing bias. All study-related personnel involved in patient care and outcome assessments remain blinded throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunosuppressive Therapy + Placebo (Placebo Comparator): Azathioprine (2.5 mg/kg/day, maximum 200 mg/day, oral) Methylprednisolone (0.5 mg/kg/day, oral, tapered over 12 weeks according to protocol) + Placebo
  Interventions: Drug: Placebo plus immunosuppression
- Immunosuppressive Therapy + Rivaroxaban (Active Comparator): Azathioprine (2.5 mg/kg/day, maximum 200 mg/day, oral) Methylprednisolone (0.5 mg/kg/day, oral, tapered over 12 weeks according to protocol), plus Rivaroxaban (20 mg/day, oral, for 12 months)
  Interventions: Drug: Rivaroxaban plus immunosupression

INTERVENTIONS:
Drug: Placebo plus immunosuppression — Participants in this arm will receive placebo plus standard immunosuppressive therapy consisting of:
  Azathioprine (2.5 mg/kg/day, maximum 200 mg/day, oral) Methylprednisolone (0.5 mg/kg/day, oral, tapered over 12 weeks according to protocol) This intervention represents the standard treatment for venous thrombosis associated with Behçet's Disease and serves as the control arm of the study.
  Arms: Immunosuppressive Therapy + Placebo
Drug: Rivaroxaban plus immunosupression — Participants in this arm will receive standard immunosuppressive therapy as described above, plus Rivaroxaban (20 mg/day, oral, for 12 months).
  This intervention aims to evaluate whether the addition of oral anticoagulation (Rivaroxaban) to immunosuppressive therapy reduces the risk of thrombotic relapse and post-thrombotic syndrome compared to immunosuppressive therapy alone.
  Arms: Immunosuppressive Therapy + Rivaroxaban

SUMMARY:
This study is a Phase III, multicenter, prospective, randomized, double-blind, placebo-controlled clinical trial investigating the treatment of lower extremity venous thrombosis associated with Behçet's Disease. The study compares the effectiveness and safety of immunosuppressive therapy alone versus immunosuppressive therapy combined with oral anticoagulation (Rivaroxaban).

DETAILED DESCRIPTION:
Behçet's Disease is a systemic inflammatory disorder that can cause vascular complications, including venous thrombosis. Although immunosuppressive therapy is the standard treatment for vascular involvement, the role of anticoagulation remains controversial. This study aims to evaluate whether adding Rivaroxaban to standard immunosuppressive treatment reduces the risk of thrombotic relapse and post-thrombotic syndrome compared to immunosuppressive therapy alone.

This study is a Phase III, multicenter, prospective, randomized, double-blind, placebo-controlled clinical trial investigating the treatment of lower extremity venous thrombosis associated with Behçet's Disease. The study compares the effectiveness and safety of immunosuppressive therapy alone versus immunosuppressive therapy combined with oral anticoagulation (Rivaroxaban).

The study will recruit patients aged 18-50 who have been diagnosed with Behçet's Disease according to International Study Group (ISG) criteria and have a newly diagnosed lower extremity venous thrombosis. Participants will be randomized (1:1) to receive either immunosuppressive therapy with Rivaroxaban or immunosuppressive therapy with a placebo. The treatment duration is 12 months, with follow-up visits at weeks 2, 4, months 2, 3, 6, 9, and 12.

The primary outcome is the rate of thrombotic relapse within 52 weeks, assessed by venous Doppler ultrasound. Secondary outcomes include the development of post-thrombotic syndrome (PTS), quality of life measures, and safety assessments, including bleeding complications.

The study is sponsored by Health Institutes of Türkiye (TÜSEB) and coordinated by Marmara University, Türkiye. Ethics approval has been obtained from Marmara University Clinical Research Ethics Committee.

For further information, please contact the study coordinators.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria to be eligible for the study:

Age between 18-50 years old. Diagnosed with Behçet's Disease according to the International Study Group (ISG) criteria.

No prior vascular involvement or no previous immunosuppressive therapy for vascular involvement.

Confirmed venous thrombosis in the lower extremity within the last 14 days before randomization.

Venous thrombosis diagnosis confirmed by:

Non-compressible venous segment in ultrasound, OR A significant (>4 mm) increase in thrombus diameter in an already abnormal segment, OR New intraluminal filling defect on venography, CT, or MR angiography.

Female participants must:

Not be pregnant or breastfeeding. Use effective contraception if of childbearing potential. Be postmenopausal (no menses for at least 1 year) or have undergone surgical sterilization.

Ability to provide written informed consent and comply with study requirements.

Exclusion Criteria:

* Participants will be excluded if they meet any of the following criteria:

Presence of any aneurysm. Chronic multisystemic disease other than Behçet's Disease. History of intolerance to Rivaroxaban. Use of immunosuppressive drugs (azathioprine, mycophenolate mofetil, cyclosporine, cyclophosphamide, TNF inhibitors, or interferon-gamma) within the last 6 months.

Prolonged corticosteroid use (>3 months) for Behçet's Disease mucocutaneous symptoms.

Prior anticoagulant therapy:

Low molecular weight heparin, fondaparinux, or unfractionated heparin for >48 hours before randomization.

More than one dose of vitamin K antagonists before randomization. Thrombectomy, vena cava filter placement, or fibrinolytic therapy for the current thrombotic episode.

Planned administration of a live vaccine within 30 days after randomization. Clinically significant acute or uncontrolled chronic diseases (e.g., cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy, or infectious diseases) that may interfere with study results.

Planned surgical procedure or significant medical condition deemed unsuitable for the study by the investigator.

History of malignancy within the last 5 years (except adequately treated basal or squamous cell carcinoma or carcinoma in situ of the cervix).

Renal impairment (Creatinine clearance <30 ml/min). Severe liver disease (e.g., acute hepatitis, active chronic hepatitis, cirrhosis, or ALT >3 times the upper limit).

Active bleeding or high bleeding risk contraindicating anticoagulant therapy. Uncontrolled hypertension (SBP >180 mmHg or DBP >110 mmHg). Severe anemia (Hemoglobin <10 mg/dL). Women who are pregnant, breastfeeding, or of childbearing potential without contraception.

Use of strong CYP3A4 inhibitors or inducers (e.g., protease inhibitors, systemic ketoconazole, rifampin, carbamazepine, phenytoin).

Participation in another experimental drug study within the last 30 days. Life expectancy of less than 3 months. History of serious infections within the last 60 days (e.g., bacterial endocarditis, tuberculosis, opportunistic infections).

Active substance or alcohol abuse or history of substance dependence within the last year.

Positive screening for Hepatitis B surface antigen, Hepatitis C antibody, or known HIV-1 infection.

Known coagulation disorders or laboratory abnormalities (e.g., DMID toxicity scale Grade 3 or higher).

History of suicidal behavior in the last 6 months or suicidal ideation (C-SSRS type 4 or 5) in the last 2 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Thrombotic Relapse at 52 Weeks | 52 weeks
  The primary outcome is the rate of thrombotic relapse within 52 weeks, assessed via lower extremity venous Doppler ultrasound.
  Thrombotic relapse is defined as:
  A new thrombotic event in a previously unaffected ipsilateral or contralateral vein.
  Re-thrombosis in a previously affected vein that was classified as well-recanalized (≥50% compressibility on Doppler ultrasound).
  Venous Doppler ultrasound assessments will be performed at baseline, months 1, 3, 6, 9, and 12.

SECONDARY OUTCOMES:
Development of Post-Thrombotic Syndrome (PTS) at 52 Weeks | 52 weeks
  The occurrence of Post-Thrombotic Syndrome (PTS) will be assessed using standardized clinical scoring systems, including:
  Villalta Scale (PTS severity assessment) Venous Clinical Severity Score (VCSS) Venous Disability Score (VDS) Venous Insufficiency Epidemiological and Economic Study Quality of Life (VEINES-QOL) PTS is defined as a Villalta score ≥5 or the presence of a venous ulcer.
Rate of Venous Recanalization at 52 Weeks | 52 weeks
  Venous recanalization will be assessed via Doppler ultrasound to evaluate the extent of clot resolution in affected veins.
  Partial or complete recanalization will be determined based on compressibility and flow characteristics.
  Measured at baseline, months 1, 3, 6, 9, and 12.
Incidence of Major and Clinically Relevant Non-Major Bleeding Events | 52 weeks
  The frequency of major bleeding (as per ISTH criteria) and clinically relevant non-major bleeding will be recorded.
  Major bleeding:
  * 2.0 g/dL hemoglobin drop
  * 2 units of red blood cell transfusion Intracranial, retroperitoneal, or fatal bleeding
  Clinically relevant non-major bleeding:
  Epistaxis >5 minutes, spontaneous hematomas >25 cm², gastrointestinal bleeding not meeting major criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Alibaz-Oner, Prof, Principal Investigator — Marmara University
Locations (2):
- Turkey (Türkiye) (2):
  - Marmara University, School of Medicine, Division of Rheumatology, Istanbul
  - Marmara University, Istanbul

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared to ensure patient confidentiality and compliance with data protection regulations